CLINICAL TRIAL: NCT04020393
Title: The Effect of Sphenopalatine Ganglion Block on the Postoperative Pain in Patients Undergoing Septorhinoplasty
Brief Title: The Effect of Sphenopalatine Ganglion Block in Patients Undergoing Septorhinoplasty
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Nazan Degirmenci, Principal Investigator, Bezmialem Vakif University
Other Study IDs: 12/232
Record Dates: First submitted 2019-07-12; First posted 2019-07-16 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Pain, Postoperative
Keywords: septorhinoplasty; sphenopalatine ganglion; postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Block group: The patients that had received Sphenopalatine ganglion block(SPGB) before the surgery
  Interventions: Procedure: SPGB
- Control Group: The patients that had not received SPBG before the surgery

INTERVENTIONS:
Procedure: SPGB — SPGB was performed by the operating surgeon using a transnasal endoscopic approach before septorhinoplasty in the Block group. The prepared solution (4 cc % 4 lidocaine and 1 cc 8 mg dexamethasone) was delivered by a Mucosal Atomization device (LMA MADgic™ Laryngo-Tracheal Mucosal Atomization Device, US). 2,5 cc of the prepared solution was given to each side of the nose.
  Groups: Block group

SUMMARY:
The investigators reviewed retrospectively the patients that had received septorhinoplasty(SRP). 42 patients were included in the study. Demographic, clinical, surgical, and follow-up data were collected from clinical case notes. The patients that had received sphenopalatine ganglion block(SPGB) before the surgery included in the Block group (n:20) and the patients that had not received SPBG before the surgery included in the Control group (n:22). The postoperative pain(POP) scores, the amount of postoperative rescue analgesics that was used, and the postoperative nausea and vomiting(PONV) scores in the first 24 hours and, mean arterial pressure (MAP), the dose of Remifentanil that was used during the operation were compared between the groups.

DETAILED DESCRIPTION:
The patients that had received SRP surgery between January-July 2019, divided into two groups according to the status of receiving SPGB before the surgery. The SPGB was done after the patient anesthetized and performed by the operating surgeon using a transnasal endoscopic approach through the posterior and over the middle turbinate tail in the pterygopalatine fossa. The patient was placed in the supine position with head extension. The prepared solution (4 cc % 4 lidocaine and 1 cc 8 mg dexamethasone) was delivered by a Mucosal Atomization device (LMA MADgic™ Laryngo-Tracheal Mucosal Atomization Device, US). 2,5 cc of the prepared solution was given to each side of the nose. The surgery was started 10 minutes after the application of SPBG, to allow sufficient time for the block to develop.

The open septorhinoplasty technique was done to all patients. The operations were done by the same two otorhinolaryngologists. Control group patients did not receive SPBG and had the surgery only. POP scores were questioned at both groups and postoperative analgesic protocols were the same.

POP was questioned by an anesthesiologist with a numeric rating scale (NRS) (0 = no pain, 10 = most severe pain) at the 30th minute(t1), 1st hour(t2), 4th hour (t3), 12th hour (t4) and 24th hours (t5) and analgesia was managed according to the NRS scores. If the NRS score was > 4, the patient was given Paracetamol 1000mg intravenously, and if the score was still >4 after 30 minutes the patient was given Tramadol 50 mg intravenously. Tramadol was used as rescue analgesia.

PONV was also evaluated. The data of nausea and vomiting were collected by direct questioning by the anesthesiologist at the same times with NRS questioning.

POP scores, the amount of postoperative rescue analgesics that was used, and PONV scores in the first 24 hours were compared between the groups.

Mean arterial pressure (MAP), and the dose of Remifentanil that was used during the operation were also compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* The patients that had received SRP
* The patients that had received SRP with SPGB
* The patients that had all the necessary information for the study in their files

Exclusion Criteria:

* The patients that had received additional surgery with SRP
* The patients whose data were absent
* The patients under the age of 18

Ages: 18 Years to 49 Years | Sex: All
Age Groups: Adult
Study Population: 42 patients that have been operated between January 2019 and July 2019 at a tertiary referral center were included in the study. The patients that had received SPBG before the surgery included in the Block group (n:20) and the patients that had not received SPBG before the surgery included in the Control group (n:22).
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Postoperative pain(POP) | 24 hour
  POP was questioned by an anesthesiologist with a numeric rating scale (NRS) (0 = no pain, 10 = most severe pain) at the 30th minute(min)(t1), 1st hour(h)(t2), 4th hour (t3), 12th hour (t4) and 24th hour (t5).
Postoperative nausea and vomiting(PONV) | 24 hour
  The data of PONV were collected by direct questioning by the anesthesiologist at the same times with POP questioning. If there is 1 min between the episodes of vomiting, each one was considered as separate episodes. Every episode of vomiting was scored as 1 point and total score was calculated after 24 hours.
The dose of rescue analgesics | 24 hour
  If the POP score was > 4, the patient was given Paracetamol 1000mg intravenously, and if the score was still >4 after 30 minutes the patient was given Tramadol 50 mg intravenously. The average dose of Paracetamol and Tramadol that were used at the first 24 hours were compared between the groups
Mean arterial pressure(MAP) | 80-240 minute
  MAP was recorded during the operation and the values were compared between the groups.
The dose of Remifentanil | 80-240 minute
  The dose of Remifentanil that was used during the operation was noted and compared between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Nazan Degirmenci, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Degirmenci N, Ozdem A, Uysal H, Sen P, Senturk E, Ozturan O, Turkoz A. The Effect of Sphenopalatine Ganglion Block on the Postoperative Pain in Patients Undergoing Septorhinoplasty. Ann Otol Rhinol Laryngol. 2020 Jul;129(7):722-726. doi: 10.1177/0003489420909417. Epub 2020 Feb 22. PMID 32090594